CLINICAL TRIAL: NCT05147155
Title: How Much Severe is the Severe Asthma of Patients Who Will be Medicated With Mepolizumab? Μeasurement of Respiratory Mechanics by Means of Impulse Oscillometry in Severe Eosinophilic Asthmatics Before and After Mepolizumab Initiation
Brief Title: Impulse Oscillometry Measurements in Severe Eosinophilic Asthmatics Before and After Anti-IL-5 Factor Initiation
Acronym: IMPOSE
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ourania Kotsiou, Assistant Professor, University of Thessaly
Other Study IDs: 15745/19-04-2021
Record Dates: First submitted 2021-06-25; First posted 2021-12-07 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Severe asthma patients: The sample will consist of 40 patients between 18 and 82 years of age with uncontrolled severe eosinophilic asthma despite receiving high dose ICS/LABA combination therapy who will receive mepolizumab, which will be administered as a 100-mg subcutaneous dose every four weeks
  Interventions: Biological: Mepolizumab
- Control group 1: Control group 1 will be a set of 50 healthy individuals matched for age and gender
- Control group 2: Control group 2 will be a set of 40 patients with severe well-controlled asthma requiring high dose ICS/LABA combination therapy from becoming uncontrolled, as previously defined, matched for age and gender.

INTERVENTIONS:
Biological: Mepolizumab — This will be a 2-year prospective study. Patients with uncontrolled severe asthma will receive mepolizumab according to standard of care and best clinical practice, which will be administered as a 100-mg subcutaneous dose every four weeks.
  Other Names: Nucala
  Groups: Severe asthma patients

SUMMARY:
Eosinophilic inflammation in the small airways of patients with severe asthma is considered to be an important marker of disease severity. In clinical trials, treatment with mepolizumab reduces exacerbation rates by almost a half along with modest improvements in symptom scores and forced expiratory volume in 1 s (FEV1) early after the first month of commencing mepolizumab treatment. However, there is an apparent discrepancy between major patient-reported outcomes and lung function that should be explored.

It has recently been reported that mepolizumab improves small airway function in severe eosinophilic asthma as detected by multiple-breath nitrogen washout test. The improvement in small airway function was seen rapidly after the first mepolizumab injection and was associated with a sustained response in the majority of patients. However, gaps in knowledge about the choice of device, gas, and standardization across systems are key issues leading the committee to conclude that multiple-breath nitrogen washout test is not ready for use as a clinical trial endpoint in asthmatics.

The investigators hypothesize that early improvement in small airway function may be a significant contributor to the therapeutic response of anti-IL-5 monoclonal antibody therapy in patients with severe uncontrolled eosinophilic asthma. The investigators speculate that SAD could be effectively evaluated using IOS. Consequently, this study could lead to novel SAD subtypes with possible clinical relevance in the context of treatment with anti-IL-5 factor. The investigators hypothesize that healthy individuals and patients with severe controlled asthma would disclose a lesser extent of SAD than patients with severe uncontrolled eosinophilic asthma with or without fixed airway obstruction.

DETAILED DESCRIPTION:
Asthma is an inflammatory condition impacting the entire bronchial tree, with small airways playing a crucial role. Small airways, defined as those less than 2 mm in diameter, are significantly involved in all stages of asthma, particularly severe cases. This region, known as the silent zone, is often linked with poor asthma control, increased severity, and a higher risk of exacerbations. Structural changes at the peribronchiolar level, such as increased stiffness due to remodeling, contribute to the disease's pathogenesis. These changes are associated with more frequent exacerbations and poorer quality of life.

Small airways account for a significant portion of airway resistance, particularly in obstructive diseases like asthma. For example, resistance in small airways can constitute up to 51% of total airway resistance in severe asthma cases. Despite their importance, measuring small airway inflammation and dysfunction remains challenging. Various tests, including spirometry and impulse oscillometry (IOS), are used, but each has limitations in detecting and evaluating small airway disease (SAD).

Methods More refined techniques like IOS are employed to better understand and treat SAD. IOS measures airway resistance and reactance during breathing without patient effort, offering a detailed analysis more sensitive to small airway changes than traditional spirometry. This technique is crucial for identifying different subtypes of SAD and is associated with asthma severity stages and control.

In clinical practice, forced oscillation technique (FOT) devices, including newer models that utilize multiple sound frequencies, are becoming popular for assessing respiratory impedance in diseases like asthma. These devices, particularly IOS, help differentiate between small and large airway obstructions and are easier to use in diverse patient groups, including the elderly and children.

Research Focus Recent studies have highlighted the effectiveness of new treatments like mepolizumab in improving small airway function in severe eosinophilic asthma. This improvement, detectable through methods like the multiple-breath nitrogen washout test, occurs quickly after treatment begins and is sustained over time. However, gaps in standardization and device choice remain challenges.

Study Objectives and Design The upcoming study will investigate early changes in respiratory mechanics using IOS in patients with severe eosinophilic asthma starting on mepolizumab. This 2-year prospective cohort study will involve 40 patients with severe asthma, matched controls for age and gender, and will assess various respiratory parameters and asthma control metrics. Measurements will be taken at multiple points to gauge the treatment's effectiveness and its impact on lung function.

Ethical Considerations The study will adhere to ethical standards, with informed consent obtained from all participants and approval from relevant ethical bodies. The goal is to enroll patients efficiently and effectively, leveraging networks of healthcare providers and educational programs to support patient recruitment and data collection.

Conclusion This research aims to enhance our understanding of SAD in severe asthma and improve treatment outcomes through innovative diagnostic techniques and targeted therapies. By focusing on the small airways, which play a significant role in asthma pathology but are challenging to study, this work could lead to more effective management strategies for those most affected by this condition.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female outpatient aged 18 to 82 years inclusive
* History of bronchial asthma for at least six months as defined by ATS criteria.
* The patients will be required to have one or more of the following objective physiological criteria: positive results on methacholine or mannitol challenge during the previous year, bronchodilator reversibility to 400 mg of inhaled Salbutamol of FEV1 ≥12% and 200ml or peak flow variability of ≥20% over two weeks.
* Diagnosis of severe asthma, defined as asthma that requires treatment with high dose inhaled corticosteroids plus a second controller and/or systemic corticosteroids to prevent it from becoming uncontrolled or that remains uncontrolled despite this therapy.
* All patients will be medicated with at least 880 μg of fluticasone propionate or the equivalent by inhalation per day and at least three months of treatment with an additional controller. Patients will be allowed to continue their anti-asthma therapy throughout the study.
* Patients should have uncontrolled asthma commencing mepolizumab treatment, based on investigator assessment, including one or both of the following:
* Poor symptom control (frequent symptoms or reliever use, activity limited by asthma, night waking due to asthma), defined as ACQ consistently ⩾1.5 or ACT<20.
* Frequent exacerbations (≥2/year) requiring oral corticosteroids, or severe exacerbations (≥1/year) requiring hospitalization or burst of systemic corticosteroids (≥3 days).
* All patients will have an eosinophil count of at least 150 cells per microliter in the peripheral blood at screening or at least 300 cells per microliter at some time during the previous year.

Exclusion Criteria:

Principal exclusion criteria:

* Diseases and health status: clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation suffering from COPD (i.e., chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* Asthmatic patients and healthy controls currently smoking or with a smoking pack history greater than 10 will be excluded.

Common exclusion criteria:

* pregnancy
* intention to become pregnant during the course of the study
* breastfeeding
* participation in another study within the 30 days preceding and during the present study
* known or suspected non-compliance, alcohol or drug abuse
* inability to follow the procedures of the study, e.g., due to language problems, psychological disorders

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will consist of 40 patients between 18 and 82 years of age with uncontrolled severe eosinophilic asthma despite receiving high-dose ICS/LABA combination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos I Gourgoulianis, Professor, Study Director — University of Thessaly
Locations (1):
- External Unit of Asthma of Respiratory Medicine Department of the University of Thessaly in Greece, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kotsiou OS, Kirgou P, Siachpazidou D, Bartziokas K, Tourlakopoulos K, Malli F, Pinaka M, Daniil Z, Gourgoulianis KI. Early benefit of mepolizumab on small airways in severe asthma: insights from the IMPOSE study. ERJ Open Res. 2025 Jun 23;11(3):00939-2024. doi: 10.1183/23120541.00939-2024. eCollection 2025 May. PMID 40551802
- Available data/document: Clinical Study Report: 10.1183/23120541.00939-2024 — https://publications.ersnet.org/content/erjor/early/2024/11/21/2312054100939-2024 — Kotsiou Ourania S., Kirgou Paraskevi, Siachpazidou Dimitra, Bartziokas Konstantinos, Tourlakopoulos Konstantinos, Malli Foteini, Pinaka Maria, Daniil Zoe, Gourgoulianis Konstantinos I. Early benefit of mepolizumab on small airways in severe asthma: insights from IMPOSE study. ERJ Open Research 2024 00939-2024; DOI: https://doi.org/10.1183/23120541.00939-2024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Started | 40 | 50 | 40
Completed | 40 | 50 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with severe uncontrolled asthma who were initiating mepolizumab treatment had significantly higher eosinophil counts, rates of early-onset asthma, allergic rhinitis, and nasal polyps compared to well-controlled asthma patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2 | Total
Number analyzed (Participants) | 40 | 50 | 40 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 40 | 30 | 100
  >=65 years | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12) | 58 (11) | 56 (14) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 35 | 24 | 86
  Male | 13 | 15 | 16 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 50 | 40 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 40 | 50 | 40 | 130
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Greece | 40 | 50 | 40 | 130
Early-onset asthma [Count of Participants; unit: Participants] | 7 | 0 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Airway Resistance at 5 Hz (R5) at Baseline (Pre-mepolizumab Initiation)
Description: Measurements of R5 at baseline (pre-mepolizumab initiation). R5 was assessed using impulse oscillometry. The values are reported in kPa/L/s and were analyzed following the guidelines of the European Respiratory Society
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.51 (0.25) | 0.39 (0.12) | 0.43 (0.16)

2. Primary Outcome: Airway Resistance at 20 Hz (R20) at Baseline
Description: Measurement of R20 at baseline - mepolizumab initiation. R20 was measured using impulse oscillometry, representing airway resistance at 20 Hz. Values are reported in kPa/L/s, and assessments were conducted according to the standards outlined by the European Respiratory Society.
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.4 (0.1) | 0.3 (0.07) | 0.3 (0.09)

3. Primary Outcome: Difference Between Airway Resistance at 5 Hz (R5) and 20 Hz (R20) at Baseline / (R5-R20) at Baseline
Description: Measurement of R5-R20 at baseline. R5-R20 represents the difference between airway resistance at 5 Hz (R5) and 20 Hz (R20), measured using impulse oscillometry. This measure reflects peripheral airway resistance. Assessments were conducted at baseline, and values are reported in kPa/L/s following guidelines from the European Respiratory Society
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.12 (0.1) | 0.05 (0.04) | 0.09 (0.08)

4. Primary Outcome: Reactance Area (AX) at Baseline
Description: Measurement of AX at baseline. AX, the area of reactance derived from impulse oscillometry, represents the elastic and inertial properties of the lungs. Measurements were taken at baseline using standard protocols. Values are reported in kPa/L and analyzed following guidelines from the European Respiratory Society.
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | 1.2 (0.8) | 0.5 (0.5) | 0.7 (0.6)

5. Primary Outcome: Resonant Frequency (Fres) at Baseline
Description: Measurement of Fres at Baseline. Fres, the resonant frequency, is the point where the reactance of the respiratory system equals zero, indicating the balance between elastic and inertial forces in the lungs. Measurements were taken at baseline using impulse oscillometry. Values are reported in Hz and analyzed following guidelines from the European Respiratory Society
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
Hz | 35 (17) | 9 (5) | 16 (7)

6. Primary Outcome: Respiratory Reactance at 5 Hz (X5) at Baseline
Description: Measurement of X5 at Baseline. X5, the respiratory reactance at 5 Hz, is a measure of the elastic properties of the lungs and the peripheral airways. It indicates how easily the lungs expand and contract during breathing. Measurements were taken at baseline using impulse oscillometry, with values expressed in kPa/L. Assessments followed European Respiratory Society guidelines. X5 is negative because the lungs store energy due to their elasticity, which results in a delayed response of airflow relative to pressure changes. This behavior is characteristic of a capacitive system, where elastic forces dominate at low frequencies. A less negative X5 means that the lung's elastic recoil is reduced, leading to decreased resistance to expansion.
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | -0.1 (0.33) | -0.08 (0.02) | -0.09 (0.04)

7. Primary Outcome: Airway Resistance at 5 Hz (R5) at Week 4.
Description: Estimate the airway resistance measured at the 5 Hz frequency (R5) after four weeks from mepolizumab initiation (only severe uncontrolled asthma patients received mepolizumab). R5 was assessed using impulse oscillometry. The values are reported in kPa/L/s and were analyzed following the guidelines of the European Respiratory Society.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.49 (0.3) | 0.3 (0.1) | 0.43 (0.16)

8. Primary Outcome: Airway Resistance at 20 Hz (R20) at Week 4.
Description: Estimate the airway resistance measured at the 20 Hz frequency (R20) after four weeks from mepolizumab initiation. R20 was measured using impulse oscillometry, representing airway resistance at 20 Hz. Values are reported in kPa/L/s, and assessments were conducted according to the standards outlined by the European Respiratory Society
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.4 (0.09) | 0.3 (0.09) | 0.3 (0.07)

9. Primary Outcome: Difference Between Airway Resistance at 5 Hz (R5) and 20 Hz (R20) at Week 4/ R5-R20 at Week 4.
Description: After four weeks of mepolizumab initiation, estimate the small airway resistance (R5- R20). R5-R20 represents the difference between airway resistance at 5 Hz (R5) and 20 Hz (R20), measured using impulse oscillometry. This measure reflects peripheral airway resistance. Assessments were conducted after 4 weeks from mepolizumab initiation, and values are reported in kPa/L/s following guidelines from the European Respiratory Society
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.10 (0.03) | 0.04 (0.03) | 0.09 (0.08)

10. Primary Outcome: Reactance Area (AX) at Week 4
Description: Estimate the AX after four weeks from mepolizumab initiation. AX, the area of reactance derived from impulse oscillometry, represents the elastic and inertial properties of the lungs. Measurements were taken at Week 4 using standard protocols. Values are reported in kPa/L and analyzed following guidelines from the European Respiratory Society.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | 0.7 (0.6) | 0.5 (0.5) | 0.7 (0.6)

11. Primary Outcome: Resonant Frequency (Fres) at Week 4.
Description: Estimate Fres after four weeks from mepolizumab initiation. Fres, the resonant frequency, is the point at which the reactance of the respiratory system equals zero, reflecting the balance between the elastic and inertial forces of the lungs. Measurements were taken at Week 4 using impulse oscillometry. Values are expressed in Hz and analyzed in accordance with European Respiratory Society guidelines.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
Hz | 17 (5) | 10 (5) | 16 (7)

12. Primary Outcome: Respiratory Reactance at 5 Hz (X5) at Week 4.
Description: Estimate X5 after four weeks from mepolizumab initiation. X5, the respiratory reactance at 5 Hz, is a measure of the elastic properties of the lungs and peripheral airways, reflecting the ability of the respiratory system to expand and contract. Measurements were taken at Week 4 using impulse oscillometry. Values are reported in kPa/L and were analyzed according to European Respiratory Society guidelines. X5 is negative because the lungs store energy due to their elasticity, which results in a delayed response of airflow relative to pressure changes. This behavior is characteristic of a capacitive system, where elastic forces dominate at low frequencies. A less negative X5 means that the lung's elastic recoil is reduced, leading to decreased resistance to expansion.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | -0.1 (0.1) | -0.08 (0.04) | -0.09 (0.04)

13. Primary Outcome: Airway Resistance at 5 Hz (R5) at Week 12
Description: Estimate the airway resistance measured at the 5 Hz frequency (R5) after 12 weeks from the mepolizumab initiation. R5 was assessed using spirometry with impulse oscillometry. The values are reported in kPa/L/s and were analyzed following the guidelines of the European Respiratory Society.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.51 (0.25) | 0.3 (0.1) | 0.43 (0.16)

14. Primary Outcome: Airway Resistance at 20 Hz (R20) at Week 12
Description: Estimate the airway resistance measured at the 20 Hz frequency (R20) after 12 weeks from mepolizumab initiation. R20 was measured using impulse oscillometry, representing airway resistance at 20 Hz. Values are reported in kPa/L/s, and assessments were conducted according to the standards outlined by the European Respiratory Society.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.4 (0.1) | 0.3 (0.09) | 0.3 (0.07)

15. Primary Outcome: Difference Between Airway Resistance at 5 Hz (R5) and 20 Hz (R20) at Week 12 / R5-R20 at Week 12
Description: Estimate small airway resistance (R5-R20) after 12 weeks from mepolizumab initiation. R5-R20 represents the difference between airway resistance at 5 Hz (R5) and 20 Hz (R20), measured using impulse oscillometry. This measure reflects peripheral airway resistance. Assessments were conducted at week 12 after mepolizuamb initiation, and values are reported in kPa/L/s following guidelines from the European Respiratory Society.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.13 (0.03) | 0.04 (0.03) | 0.09 (0.08)

16. Primary Outcome: Reactance Area (AX) at Week 12
Description: Estimate the AX after 12 weeks from mepolizumab initiation. AX, the area of reactance derived from impulse oscillometry, represents the elastic and inertial properties of the lungs. Measurements were taken at Week 12 using standard protocols. Values are reported in kPa/L and analyzed following guidelines from the European Respiratory Society.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | 0.7 (0.5) | 0.5 (0.5) | 0.7 (0.6)

17. Primary Outcome: Resonant Frequency (Fres) at Week 12
Description: Estimate Fres after12 weeks from mepolizumab initiation. Fres, the resonant frequency, is the point at which the reactance of the respiratory system equals zero, reflecting the balance between the elastic and inertial forces of the lungs. Measurements were taken at Week 4 using impulse oscillometry. Values are expressed in Hz and analyzed in accordance with European Respiratory Society guidelines.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
Hz | 17 (6) | 10 (5) | 16 (7)

18. Primary Outcome: Respiratory Reactance at 5 Hz (X5) at Week 12
Description: Estimate X5 after 12 weeks from mepolizumab initiation. X5, the respiratory reactance at 5 Hz, measures the elastic properties of the lungs and peripheral airways, reflecting the ability of the respiratory system to expand and contract. Measurements were taken at Week 12 using impulse oscillometry. Values are reported in kPa/L and analyzed according to European Respiratory Society guidelines. X5 is negative because the lungs store energy due to their elasticity, which results in a delayed response of airflow relative to pressure changes. This behavior is characteristic of a capacitive system, where elastic forces dominate at low frequencies. A less negative X5 means that the lung's elastic recoil is reduced, leading to decreased resistance to expansion.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | -0.1 (0.1) | -0.08 (0.04) | -0.09 (0.04)

19. Primary Outcome: Airway Resistance at 5 Hz (R5) at Week 26.
Description: Estimate the airway resistance measured at the 5 Hz frequency (R5) after 26 weeks from the initiation of mepolizumab. R5 was assessed using spirometry with impulse oscillometry. The values are reported in kPa/L/s and were analyzed following the guidelines of the European Respiratory Society.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.41 (0.1) | 0.3 (0.1) | 0.43 (0.16)

20. Primary Outcome: Airway Resistance at 20 Hz (R20) at Week 26.
Description: Estimate the airway resistance measured at the 20 Hz frequency (R20) after 26 weeks from mepolizumab initiation. R20 was measured using impulse oscillometry, representing airway resistance at 20 Hz. Values are reported in kPa/L/s, and assessments were conducted according to the standards outlined by the European Respiratory Society.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.4 (0.1) | 0.3 (0.09) | 0.3 (0.07)

21. Primary Outcome: Difference Between Airway Resistance at 5 Hz (R5) and 20 Hz (R20) at Week 26 / R5-R20 at Week 26.
Description: Estimate the small airway resistance (R5-R20) after 26 weeks from mepolizumab initiation. R5-R20 represents the difference between airway resistance at 5 Hz (R5) and 20 Hz (R20), measured using impulse oscillometry. This measure reflects peripheral airway resistance. Assessments were conducted at Week 26 after mepolizumab initiation, and values are reported in kPa/L/s following guidelines from the European Respiratory Society
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kPa/L/s
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L/s | 0.03 (0.03) | 0.04 (0.03) | 0.09 (0.08)

22. Primary Outcome: Reactance Area (AX) at Week 26.
Description: Estimate AX after 26 weeks from mepolizumab initiation. AX, the area of reactance derived from impulse oscillometry, represents the elastic and inertial properties of the lungs. Measurements were taken at Week 26 using standard protocols. Values are reported in kPa/L and analyzed following guidelines from the European Respiratory Society.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | 0.6 (0.5) | 0.5 (0.5) | 0.7 (0.6)

23. Primary Outcome: Resonant Frequency (Fres) at Week 26.
Description: Estimate Fres after 26 weeks from mepolizumab initiation. Fres, the resonant frequency, is the point at which the reactance of the respiratory system equals zero, reflecting the balance between the elastic and inertial forces of the lungs. Measurements were taken at Week 26 using impulse oscillometry. Values are expressed in Hz and analyzed in accordance with European Respiratory Society guidelines.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: Hz
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
Hz | 17 (6) | 10 (5) | 16 (7)

24. Primary Outcome: Respiratory Reactance at 5 Hz (X5) at Week 26.
Description: Estimate X5 after 26 weeks from mepolizumab initiation. X5, the respiratory reactance at 5 Hz, reflects the elastic properties of the lungs and peripheral airways, indicating the ability of the respiratory system to expand and contract. Measurements were taken at Week 26 using impulse oscillometry. Values are reported in kPa/L and were analyzed following European Respiratory Society guidelines. X5 is negative because the lungs store energy due to their elasticity, which results in a delayed response of airflow relative to pressure changes. This behavior is characteristic of a capacitive system, where elastic forces dominate at low frequencies. A less negative X5 means that the lung's elastic recoil is reduced, leading to decreased resistance to expansion.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: kPa/L
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
Number analyzed (Participants) | 40 | 50 | 40
kPa/L | -0.08 (0.1) | -0.08 (0.04) | -0.09 (0.04)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for a period of 6 months following mepolizumab initiation.
Description: The definitions of adverse events and serious adverse events used to collect adverse event information were consistent with the ClinicalTrials.gov definitions. No differences were noted.
Arm/Group | Severe Asthma Patients | Control Group 1 | Control Group 2
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/50 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/50 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/50 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT05147155/Prot_SAP_000.pdf